CLINICAL TRIAL: NCT04690621
Title: Cross-sectional Examination of the Reliability of Oral Implants
Acronym: PeriX2012
Status: Completed | Type: Observational
Sponsor: German Association of Oral Implantology e. V. (Other)
Responsible Party: Sponsor
Other Study IDs: GermanAOI2012
Record Dates: First submitted 2020-12-20; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2012-06

CONDITIONS: Periimplantitis
Keywords: peri-implant disease prevalence incidence tolerance titanium
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Aim of the multi centrical, cross-sectional study is the registration of the prevalence and incidence of mucositis and periimplantitis.

DETAILED DESCRIPTION:
Aim of the multi centrical, cross-sectional study is the registration of the prevalence and incidence of mucositis and periimplantitis. Additional clinical examination of the tolerance of titanium using cytosine analysis of periimplant sulcus smear and of blood lymphocytes on titanium plates in vitro. In total 10 centers will examine clinical, genetic and microbiological parameters in 200 patients during 12 months.

Study hypothesis: The incidence of mucositis and periimplantitis during a time period of 10 years in patients is less than 30%

ELIGIBILITY:
Inclusion Criteria:

* Patients with oral implants inserted after 01.04.2002
* Periodical recall

Exclusion Criteria:

* No other titanium implants inside the body

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with oral implants inserted after 01.04.2002
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2012-07-01 (Actual); Primary Completion 2013-02-20 (Actual); Study Completion 2013-08-07 (Actual)

PRIMARY OUTCOMES:
IL-1ß | 6 month
  Interleucin 1 beta in peripheral blood

SECONDARY OUTCOMES:
MMP-8 | 6 month
  Metallomatrixproteinase-8 in Periodontal Sulcus Fluid
BOP | 6 months
  Bleeding on probing
PD | 6 months
  Probing Depth

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Iglhaut, DDS, PhD, Principal Investigator — Academy Member
Locations (1):
- Gerhard Iglhaut, Memmingen, Germany

REFERENCES:
- See also: German Association of Oral Implantology — https://www.dginet.de

DOCUMENTS (2):
  • Study Protocol (2011-12-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT04690621/Prot_000.pdf
  • Informed Consent Form (2011-12-23): https://cdn.clinicaltrials.gov/large-docs/21/NCT04690621/ICF_001.pdf